CLINICAL TRIAL: NCT05624502
Title: Mprovement in Postoperative Pain Outcome: Pain Registry
Brief Title: Improvement in Postoperative Pain Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, SALAH EL-TALLAWY, Professor and Consultant - Anesthesia and Pain Management, King Saud University
Other Study IDs: 18/0443/IRB
Record Dates: First submitted 2022-11-13; First posted 2022-11-22 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Acute Post Operative Pain
Keywords: acute postoperative pain; orthopedic surgery; general surgery; obs/gyn surgery; Neurosurgery; Bariatric surgery; Thoracic surgery; opioids; NSAIDs; Regional analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study project aims at improving postoperative pain outcomes by evaluating the current status of postoperative pain managements in the institution. Then the investigators will compare the results by internal and external benchmarking. Then they will suggest recommendations to improve the current situation of postoperative pain management.

DETAILED DESCRIPTION:
At least half of the patients suffer from moderate to severe post-operative pain. The price of poorly managed pain is high: pain impedes recovery, causes suffering and prolongs the hospital stay. PAIN OUT provides tools for measurement, feedback and benchmarking of pain treatment quality in order to improve patient care. A research project that aims at improving postoperative pain treatment outcomes by evaluating the current status of postoperative pain managements in our institution. Then the investigators compare the results by internal and external benchmarking. Then suggest recommendations to improve the current situation of postoperative pain management.

parameters include" Patient's data Pain assessments by using the visual analogue score of 11 point (from "0" no pain - "10" worst pain) will be evaluated as the following: Worst pain since surgery, Least pain since surgery, Pain score at rest. Pain score during movements in bed, Pain score during deep breathing and coughing, How often the severe pain since surgery (%), Does the pain interfere with sleeping pattern, and the side effects.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative patients during the first 24 hours of surgery (day 1)
* Male and Females
* Adults

Exclusion Criteria:

* Patient refusal
* Drug abusers and addicts
* Major significant systemic diseases
* Language barriers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute postoperative pain patients after different surgical procedures
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative pain scores | first 3 days postoperative
  using visual analogue scale (VAS) for pain assessment of 11 points (from "0" no pain to "10" worst pain
time in severe pain | during the first 24 hours
  duration of time spent in severe pain after surgery
dynamic and static pain | during the first 24 hours
  Pain scores or rest and during movements

SECONDARY OUTCOMES:
worst and least pain | during the first 24 hours
  The highest and lowest pain scores during the first 24 hours
time to first request of analgesia | during the first 24 hours
  the time from the recovery to the first request of postoperative analgesia
total analgesic consumption | during the first 24 hours
  total consumption of opioids / non-opioids during the first 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Salah N. El-Tallawy, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No